CLINICAL TRIAL: NCT03638297
Title: PD-1 Antibody Combined With COX Inhibitor in MSI-H/dMMR or High TMB Colorectal Cancer: a Single Arm Phase II Study
Brief Title: PD-1 Antibody Combined With COX Inhibitor in MSI-H/dMMR or High TMB Colorectal Cancer
Acronym: PCOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU13
Record Dates: First submitted 2018-08-17; First posted 2018-08-20 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
Keywords: MSI-H; dMMR; PD-1 antibody; COX inhibitor; tumor mutation burden
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cyclooxygenase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody + cox inhibitor (Experimental): BAT1306 + aspirin(celebrex when there is contraindication to aspirin) on day 1-21 every three weeks
  Interventions: Drug: PD-1 antibody + cox inhibitor

INTERVENTIONS:
Drug: PD-1 antibody + cox inhibitor — BAT1306 100mg /pembrolizumab 200mg on day 1 + aspirin 200mg oral (celebrex 400mg oral when there is contraindication to aspirin) on day 1-21 every three weeks
  Contraindication to aspirin :
  Allergic or intolerance to aspirin; With peptic ulcers; With hemophilia or other bleeding tendencies; Have the gentic disease glucose-6 phosphate dehydrogenase deficiency.

SUMMARY:
PD-1(programmed death protein 1)antibody has been to approved in patients with MSI-H/dMMR advanced cancer and has achieved significant efficacy. It is reported that the objective response rate of Pembrolizumab and Nivolumab are 40% and 31.1% in MSI-H/dMMR (microsatellite instability-high/deficiency mismatch repair )colorectal cancer. What's more, most of the patients who had response for PD-1 antibody achieved a long duration of disease control. However, not all patients with MSI-H/dMMR was sensitive to PD-1 antibody despite it is a biomarker for PD-1 antibody treatment. There were about 50-60% of patients with MSI-H/dMMR were insensitive and we don't know why. What's more, it's reported that tumor mutation burden (TMB) may be another biomarker of response to PD-1 therapy. COX (cyclooxygenase)inhibitor has been proved to prevent adenomas in colorectal and it is safe for most of the patients. Preclinical models also showed that COX inhibitor could act with PD-1 antibody in mice and control disease progress. So, this study aims to evaluated efficacy and safety of combination of PD-1 antibody and COX inhibitor in patients with MSI-H/dMMR or high tumor mutation burden colorectal cancer.

DETAILED DESCRIPTION:
This is a single arm, phase two study. Eligible patients with advanced MSI-H/dMMR colorectal cancer were assigned to receive BAT1306 plus COX inhibitor. All patients will receive the study regimen every 3 weeks. Chest/abdomen/pelvic CT with IV contrast will be performed to assess clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent; able to comply with study and/or follow- up procedures;
2. Age:18-75 years old;
3. Histological or cytological documentation of colorectal cancer;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. There must be documentation by CT scan, MRI, or intraoperative palpation that tumor is unresectable;
6. Have had at least one lines of chemotherapy fail or refuse to receive chemotherapy;
7. Histologically confirmed metastatic or primary colorectal cancer as dMMR/MSI-H or whole exon sequence confirmed tumor mutation burden higher than 1000;
8. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment: Hemoglobin (Hb) ≥ 90g/ L, absolute neutrophil count (ANC) ≥ 1.5×109/ L, platelet count ≥ 100×109/ L; Total bilirubin ≤ 1.5×the upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 ×ULN; Serum creatinine ≤1.5×the ULN.

Exclusion Criteria:

1. Previous treatment with other therapy targeting T-cell costimulation or immune checkpoint pathways;
2. Active, known, or suspected autoimmune disease (except for type 1 diabetes mellitus, residual hypothyroidism due to autoimmune condition requiring only hormone replacement, or conditions not expected to recur in the absence of an external trigger);
3. A previous cancer active within the previous 5 years;
4. Subjects with known allergy to the study drugs or to any of its excipients;
5. Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment;
6. Heart failure grade III/IV (NYHA-classification);
7. Patients with active infection within 1 week before enrollment (infection caused by fever above 38 °C);
8. Patients with severe lung disease (interstitial pneumonia, pulmonary fibrosis, severe emphysema);
9. Patients with active gastrointestinal bleeding;
10. Patients with serious complications (intestinal obstruction, renal insufficiency, hepatic insufficiency, cerebrovascular disorders);
11. Psychiatric disease or a history of central nervous system disease that affects clinical treatment;
12. Receive other anti-tumor treatments (including anti-tumor immunotherapy, interventional therapy and intra-serosal injection of anti-tumor drugs) or participate in other interventional clinical trials within two weeks before enrollment;
13. Breast- feeding or pregnant women;
14. Lack of effective contraception;
15. The investigator determined that the patient was not eligible for this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 months
  CR(complete response) + PR (partial response)rate will be assessed according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Time measured from the day of treatment to the date of first documented progression, or death from any cause.
Overall survival time | 5 years
  Estimated from the date of treatment to death from any cause.
disease control rate | 6 months
  CR + PR + SD(stable disease) rate will be assessed according to the RECIST version 1.1 guidelines.
Toxicity assessed using the NCI common toxicity criteria, version 4.0. | 2 years
  The grade of toxicity will be assessed using the NCI common toxicity criteria, version 4.0.
duration of response | 2 years
  Time measured from the day of first documented PR or CR to the date of first documented progression, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (2):
- China (2):
  - Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong

REFERENCES:
- [Derived] Wu Z, Zhang Y, Cheng Y, Li J, Li F, Wang C, Shi L, Qin G, Zhan W, Cai Y, Xie X, Ling J, Hu H, Zhang J, Deng Y. PD-1 blockade plus COX inhibitors in dMMR metastatic colorectal cancer: Clinical, genomic, and immunologic analyses from the PCOX trial. Med. 2024 Aug 9;5(8):998-1015.e6. doi: 10.1016/j.medj.2024.05.002. Epub 2024 May 24. PMID 38795703